CLINICAL TRIAL: NCT06778525
Title: The Effect of Rehabilitative Games With SmartPose Practice on Upper Extremity Recovery in Ischemic Stroke Patients
Brief Title: The Effect of Rehabilitative Games With SmartPose on Upper Extremity Recovery in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Cilen Tavsanoglu, Physiotherapist, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Msc thesis
Record Dates: First submitted 2025-01-11; First posted 2025-01-16 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-06

CONDITIONS: Stroke, Ischemic; Smartpose; Telerehabilitation
Keywords: Rehabilitation; Stroke; Exergaming; Upper Extremity
MeSH Terms: conditions — Ischemic Stroke; Stroke | interventions — Exercise; Rehabilitation; Exergaming

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): A one-hour exercise protocol will be administered in this group, consisting of 30 minutes of conventional exercises and 30 minutes of Smartpose exercises.
  Interventions: Other: Exercise; Other: SmartPose
- Control (Active Comparator): A one-hour conventional exercise program will be administered to this group.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Personalized neuromuscular exercises, according to the patient's specific needs.
  Other Names: Rehabilitation
Other: SmartPose — Virtual reality application containing rehabilitative games developed for individuals in need of exercise.
  Other Names: Exergame; Virtual Reality
  Arms: Experimental Group

SUMMARY:
The goal of this clinical trial is to investigate the effects of SmartPose games on upper extremity motor, functional, and sensory recovery in patients with stroke. The main question it aims to answer is:

* Does the use of rehabilitative games with the SmartPose application work to treat upper extremity motor, functional, and sensory recovery in stroke patients?

Researchers will compare the experimental group with the control group, which receives only conventional exercises with proven effectiveness, to determine whether SmartPose has an effect on upper extremity motor, functional, and sensory recovery in stroke patients.

The experimental group will receive 30 minutes of neuromuscular therapy and 30 minutes of SmartPose, 3 times a week for 8 weeks.

The control group will receive 60 minutes of neuromuscular therapy, 3 times a week for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Mini Mental State Examination score ≥ 24
* Age between 35 and 75 years
* Medical condition sufficiently stable to allow participation in active rehabilitation
* Brunnstrom Upper Extremity Stage ≥ 3
* Minimum sixth week post-stroke
* Ability to perform shoulder abduction and flexion against gravity with a minimum of 20°

Exclusion Criteria:

* Presence of secondary impairments affecting upper extremity movement
* Modified Ashworth Scale score of 4 or 5
* Inability to maintain independent sitting balance
* Visual impairment or loss that prevents the perception of visual materials

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2025-01-11 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
The Fugl-Meyer Assessment of Motor Recovery after Stroke - Upper Limb | Baseline and 8 weeks
  Fugl-Meyer is the first measure developed to quantitatively assess sensorimotor recovery after stroke. In our study, to evaluate total sensorimotor recovery, we used the motor function section of this assessment, which consists of 33 items and a total of 66 points, and the sections on sensation, passive joint movement, and joint pain, which have a total of 60 points. Higher scores reflect better motor function recovery.
Frenchay Arm Test | Baseline and 8 weeks
  FAT assesses motor control and hand skills in patients with functional loss in the upper extremity following neurological impairment. The test consists of 5 items and takes a total of 3 minutes. Each item is scored as successful (1 point) or unsuccessful (0 points). It is evaluated on a total of 5 points. Higher scores reflect better motor control.

SECONDARY OUTCOMES:
Modified Ashworth Scale | Baseline and 8 weeks
  MAS is a scale developed to assess muscle tone by determining the resistance exhibited against passive movement throughout the range of motion in the joint, and its validity has been proven in cases of stroke. The Modified Ashworth Scale (MAS) consists of six categories: 0, 1, 1+, 2, 3, and 4 (with the addition of 1+). Scoring is based on the resistance felt during passive movement of the joint, where 0 indicates no increase in muscle tone and 4 indicates a rigid joint. Lower scores reflect a lower degree of spasticity.
Brunnstrom Stages of Stroke Recovery | Baseline and 8 weeks
  Brunnstrom is an approach that can be used both as a treatment approach and to assess body functions in cases of stroke. The Brunnstrom staging system has created a common language in the rehabilitation process. Higher stages indicate closer approximation to normal motor function.
Box and Block Test | Baseline and 8 weeks
  BBT is a measure that evaluates manual dexterity based on performance. The patient was asked to move as many cubes as possible from the box in front of them to the other box next to them using the affected extremity for 60 seconds. A higher number of transferred cubes indicates better hand performance.
Functional Independence Measure | Baseline and 8 weeks
  The FIM is used to assess patients' functional status and level of independence. The test consists of two sections; motor skills and cognitive skills. Scores range from 18, indicating complete dependence, to 126, indicating full independence.
Stroke Specific Quality of Life Scale | Baseline and 8 weeks
  The Stroke-Specific Quality of Life Scale was developed to assess quality of life parameters in stroke patients. The scale consists of a total of 48 items and 8 subscales. The items of the Stroke-Specific Quality of Life Scale are rated on a 5-point scale ranging from 1 to 5. The response options are scored as '1 = strongly agree, 2 = partially agree, 3 = neutral, 4 = partially disagree, and 5 = strongly disagree.' For some items, the response options are scored as '1 = could not do at all, 2 = had great difficulty, 3 = had some difficulty, 4 = had little difficulty, and 5 = no difficulty.' Higher total scores indicate better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University-Cerrahpasa, Faculty of Health Science, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided